CLINICAL TRIAL: NCT07104903
Title: Risk Factor Assessment for Surgical Site Infection After Colorectal Cancer Surgery
Brief Title: Risk Factor Assessment for the Development of Surgical Site Infection in Patients Undergoing Colorectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Oncology Institute of Vojvodina (Other Government)
Responsible Party: Principal Investigator, Nora Mihalek, Dr, Oncology Institute of Vojvodina
Other Study IDs: 4/24/3-5228/2-9
Record Dates: First submitted 2025-07-28; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Surgical Site Infections; Colorectal Cancer
MeSH Terms: conditions — Surgical Wound Infection; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection from medical records — Data are collected from the information system and medical records, including demographic characteristics, presence of surgical site infection, comorbidities, data regarding neoadjuvant oncological therapy, preoperative laboratory findings, type and duration of surgical intervention, perioperative complications, and SENIC and NNIS scores are calculated.

SUMMARY:
Surgical site infection (SSI) is a common complication following colorectal cancer (CRC) surgery and represents a significant cause of slower postoperative recovery and prolonged hospital stay. Therefore, this study aims to determine which risk factors contribute most to SSI development, and to assess the effectiveness of SENIC and NNIS scores in evaluating SSI risk after CRC surgery.

This retrospective observational cohort study is conducted at the Oncology Institute of Vojvodina. Sixty-two patients are included, undergoing elective CRC surgery between 03.06.2024. and 31.10.2024. Data are collected from the information system and medical records, including demographic characteristics, presence of SSI, comorbidities, data regarding neoadjuvant oncological therapy, preoperative laboratory findings, type and duration of surgical intervention, perioperative complications, and SENIC and NNIS scores are calculated.

The study is supported by a Collegium Talentum scholarship from the Ministry of Human Capacities (Hungarian Government), for the 2024/2025 academic year (recipient Nora Mihalek, MD).

Contact: Nora Mihalek, MD Oncology Institute of Vojvodina, Department for Anesthesiology with Reanimatology, Sremska Kamenica, Serbia; University of Novi Sad, Faculty of Medicine, Novi Sad, Serbia

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (˃ 18 years of age)
* ASA III clinical status
* Patients undergoing radical surgical treatment of colorectal cancer

Exclusion Criteria:

- Patients undergoing palliative surgical treatment of colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective radical colorectal cancer surgery in the period between 03.06.2024. and 31.10.2024. in the Oncology Institute of Vojvodina.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infection | During hospital stay (assessed up to 15 days)
  Data collected from medical records and information system

SECONDARY OUTCOMES:
Incidence of particular risk factors for the development of surgical site infection (diabetes mellitus, anaemia, neoadjuvant chemotherapy, neoadjuvant radiotherapy) | Baseline
Incidence of particular risk factors for the development of surgical site infection (red blood cell transfusion, length of intervention > 3 hours, contaminated wound, ClassIntra classification, stoma formation) | Perioperative/Periprocedural
Study on the Efficacy of Nosocomial Infection Control (SENIC) score | Baseline
  Maximal value: 4; Minimal value: 0 (higher score indicates worse outcome)
National Nosocomial Infection Surveillance (NNIS) score | Baseline
  Maximal value: 3; Minimal value: 0 (higher score indicates worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Vojvodina, Kamenitz, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No